CLINICAL TRIAL: NCT02238275
Title: Post-Marketing Surveillance Study Micardis® Plus
Brief Title: Post-Marketing Surveillance Study of Micardis® Plus in Patients With Hypertension
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 502.390
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with hypertension
  Interventions: Drug: Micardis® plus

INTERVENTIONS:
Drug: Micardis® plus

SUMMARY:
Study to evaluate efficacy and tolerability of Micardis® plus under usual daily-practice prescribing-conditions

ELIGIBILITY:
Inclusion Criteria:

* Adult (Age >= 18 years) males and females for whom a medical antihypertensive therapy is indicated

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with hypertension
Sampling Method: Non-Probability Sample
Enrollment: 8135 (Actual)
Dates: Start 2002-06; Primary Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in morning blood pressure | Baseline, after 6 weeks
Change from baseline in classification of blood pressure | Baseline, after 6 weeks
  according to Word Health Organisation - Isolated systolic hypertension (WHO-ISH) - definition of 'Deutsche Hochdruckliga'

SECONDARY OUTCOMES:
Number of patients with adverse drug reactions | up to 6 weeks
Assessment of efficacy by investigator on 5-point scale | after 6 weeks
Assessment of tolerability by investigator on a 5-point scale | after 6 weeks
Change from baseline in heart rate | Baseline, after 6 weeks